CLINICAL TRIAL: NCT03795870
Title: The Effect of Blenderized Tube Feeding on Enteral Nutrition Tolerance and the Gut Microbiome: A Pilot Study
Brief Title: Enteral Nutrition Tolerance and the Gut Microbiome Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Manpreet S. Mundi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 18-004416
Record Dates: First submitted 2018-12-10; First posted 2019-01-08 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Enteral Feeding Intolerance
Keywords: Home Enteral Nutrition; Gut Microbiome; Blenderized Tube Feeds

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization list will be generated using http://www.randomization.com and the investigator team will be blinded at enrollment using supplement codes. A designated study coordinator will hold the randomization codes and the codes will be revealed to the investigators only after the statistical analysis is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polymeric Tube Feeds (Active Comparator): This arm will be receiving Polymeric Tube Feeds as a part of the regular HEN Protocol.
  Interventions: Dietary Supplement: Polymeric Tube Feeds
- Blenderized Tube Feeds (Active Comparator): This arm will be receiving Blenderized tube feeds as a part of the regular HEN Protocol.
  Interventions: Dietary Supplement: Blenderized Tube Feeds

INTERVENTIONS:
Dietary Supplement: Polymeric Tube Feeds — Polymeric tube feeds will be given to HEN patients to assess the percentage of goal calories provided in comparison with blenderized tube feeds
  Arms: Polymeric Tube Feeds
Dietary Supplement: Blenderized Tube Feeds — Blenderized tube feeds will be given to HEN patients to assess the percentage of goal calories provided in comparison with polymeric tube feeds
  Arms: Blenderized Tube Feeds

SUMMARY:
The current study will enroll patients who are going to require enteral nutrition support for at least 4 weeks and randomize them to standard polymeric formulas or blenderized tube feeding. They will be asked to fill out a questionnaire about their tolerance of enteral feeds. They will also be asked to provide stool samples before enrollment and after 4-6 weeks.

The study is trying to assess whether the use of whole food in blenderized tube feeding will be better tolerated and also lead to greater diversity of microbiome.

DETAILED DESCRIPTION:
Malnutrition remains highly prevalent in both acute and chronic diseases, leading to longer hospital length of stay, greater risk of hospital readmission, and overall increase in morbidity and mortality. Over the last few decades, studies have continued to reveal significant clinical benefit from nutrition support, including reduction in complications and length of stay, maintenance of gastrointestinal integrity, and overall improvement in clinical outcomes and mortality. Despite high prevalence of Home Enteral Nutrition(HEN), patients continue to struggle with intolerance of tube feeds leading to chronic underfeeding and weight loss. Current guidelines recommend using standard polymeric formula or high-protein standard formula in the hospitalized patient requiring EN and also recommend against routine use of formulas designed to be immune-modulatory, elemental/semi-elemental, disease-specific (diabetes), and organ-specific (hepatic, renal, pulmonary).

Blenderized Tube Feeding(BTF) offers a number of advantages to standard polymeric formula including being able to modify the macro-nutrient and fiber content based on patient preference. BTF use has also been increasing significantly in the past few years.

The gut microbiome, or gut host environment, consists of approximately 10 thousand cells and has been the subject of much interest as it relates to gastrointestinal homeostasis. Our aim therefore is to (1) characterize the structure and dynamics of complex microbial communities using 16S rRNA- encoding gene sequences; (2) determine how they change with EN and; (3) how they may be correlated with tolerance of EN.

A total of fifty subjects who are willing to participate in current trial and who meet eligibility will be recruited from the Mayo Clinic HEN program. Suitable subjects will be identified when they present at the initial HEN visit prior to undergoing enteral tube placement.

Written informed consent will be obtained from all individuals who participate in the study. The principal investigator or member of study team meet with each participant, review the consent form in detail and confirm the subject's understanding of the study. The study team will answer all questions posed by the participants and when convinced that the subject verbally demonstrates understanding of the protocol, they will obtain a signed consent. Only designated staff members are authorized to obtain informed consent.

At the pre-enteral tube visit, subjects will complete a gastrointestinal quality of life (QoL) questionnaire which will form the baseline assessment for symptoms and functional status. Body composition will be measured using Bio-impedance analysis (BIA; InBody™). A stool specimen will be obtained for analysis of the gut microbiome at baseline. Baseline clinical data such as current medical problems will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects who are above 18 years of age, who present to Mayo Clinic HEN program for initial evaluation prior to enteral tube placement
2. Require enteral nutrition support for at least 4-6 weeks from enrollment

Exclusion Criteria:

1. Patients with type 1 or 2 diabetes will be excluded due to the known pre-existing changes in the gut microbiome in this population.
2. Patients who have had exposure to probiotics, prebiotics or antibiotics in the preceding 4 weeks will be excluded.
3. Known allergy or intolerance to study products will be excluded.
4. Patients on parenteral nutrition will be excluded.
5. If oral feeding accounts for >25% of daily caloric intake.
6. Presence of entero-cutaneous fistula
7. Patients with short bowel syndrome will be excluded.
8. Patients who have had bariatric surgery or other alteration of GI tract will be excluded.
9. Hematologic malignancy with absolute neutrophil count < 500/mm3
10. History of renal or liver transplant or on transplant list.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Percentage of goal calories provided | 4-6 weeks

SECONDARY OUTCOMES:
Gut microbiome | 1 week, 4-6 weeks
  A stool specimen will be collected to assess the composition of the gut microbiome at baseline and at the follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet S Mundi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No